CLINICAL TRIAL: NCT05507112
Title: The Therapeutic and Prognostic Implications of Tumor Immune Microenvironment in The Neoadjuvant Immunotherapy Combined With Chemoradiotherapy for Rectal Cancer
Brief Title: TIME in Immunotherapy Combined With nCRT for Rectal Cancer
Acronym: TIMENT-R
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH_TIMENT-R
Record Dates: First submitted 2022-07-17; First posted 2022-08-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-07

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Rectal Cancer; Immunotherapy; neoadjuvant therapy; Tumor Immune Microenvironment
MeSH Terms: conditions — Rectal Neoplasms | interventions — Immune Checkpoint Inhibitors; tislelizumab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemoradiotherapy plus PD-1 inhibitor (Experimental): Capecitabine 1650mg/m2 is given 5 days a week in parallel with radiotherapy 45 to 50 Gy during 5 consecutive weeks.
  Tislelizumab is given on day 1 of week 2, 5 and 8 at 200 mg i.v. 8-12 weeks after completion of radiation therapy, patients undergo total mesorectal excision (TME).
  Interventions: Drug: PD-1 inhibitor; Drug: Capecitabine; Radiation: Long-course radiation therapy
- Neoadjuvant chemoradiotherapy (Active Comparator): Capecitabine 1650mg/m2 is given 5 days a week in parallel with radiotherapy 45 to 50 Gy during 5 consecutive weeks.
  8-12 weeks after completion of radiation therapy, patients undergo total mesorectal excision (TME).
  Interventions: Drug: Capecitabine; Radiation: Long-course radiation therapy

INTERVENTIONS:
Drug: PD-1 inhibitor — Tislelizumab (3 cycles): 200mg i.v. q3w on day 1 of each cycle, and starting from the second week after the start of radiotherapy
  Other Names: Tislelizumab
  Arms: Neoadjuvant chemoradiotherapy plus PD-1 inhibitor
Drug: Capecitabine — Capecitabine 1650mg/m2/d orally twice-daily, 5 days a week for a total of 5 weeks.
  Other Names: Xeloda
Radiation: Long-course radiation therapy — 45-50 Gy/day, 5 days a week for a total of 5 weeks.

SUMMARY:
This is an open-label, prospective phase II clinical trial to evaluate the therapeutic and prognostic implications of tumor immune microenvironment in the neoadjuvant immunotherapy combined with chemoradiotherapy for patients with rectal cancer. A total of 100 patients will be enrolled in this trial. The primary end point is the rate of pathological complete response (pCR). The long-term prognosis and adverse effects will also be evaluated and analyzed.

DETAILED DESCRIPTION:
Objectives:

1. To clarify the efficacy and safety of combined therapy for locally advanced rectal cancer (LARC) patients and verify the efficacy and safety of neoadjuvant immunotherapy for dMMR/MSI-H LARC patients.
2. To clarify the effect of nCRT on TIME for rectal cancer, and the further effect of adding Immunotherapy.
3. To verify the feasibility of predicting the efficacy of combined therapy by the infiltration level of CD8+ PD1+ TILs in tumor tissue before treatment in pMMR/MSS LARC patients and explore the comprehensive prediction index of the efficacy of combined therapy for LARC patients.
4. To clarify the potential mechanism of immune response or immune escape to neoadjuvant immunotherapy for LARC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤75 years on the day of signing informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
3. Histologically proven rectal adenocarcinoma.
4. <12 cm from anal verge.
5. Clinical stage of T3/T4 or N positive and M0
6. No previous chemotherapy, radiotherapy, immunotherapy or surgical treatment
7. No immune system disease (e. g. systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), systemic vasculitis, scleroderma, mixed connective tissue disease, dermatomyositis (DM), hyperthyroidism, hypothyroidism, ulcerative colitis (UC), autoimmune hemolytic anemia (AIHA) or human immunodeficiency virus (HIV) infection.
8. Adequate hepatic and renal function to chemoradiotherapy, immunotherapy and surgery.
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Allergic to any component of chemotherapy or immunotherapy;
2. Patients with multiple primary colorectal cancer;
3. Other malignant tumors within 5 years, except for adequately treated cervical carcinoma in situ or cutaneous basal cell carcinoma, or basically controlled localized prostate cancer or surgically excised ductal carcinoma in situ of breast;
4. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, or other conditions requiring emergency surgical resection;
5. Prior or planed organ/bone marrow transplant
6. Patients who receive systemic steroid therapy or immunosuppressive agents within 30 days before enrollment in the study;
7. Pregnant or lactating women
8. Patients with a history of severe mental illness or being unable to comply with the research protocols.
9. Patients who have contraindications to chemoradiotherapy, immunotherapy or surgery.
10. Patients who have any other conditions that investigator judges unsuitable to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rates | 1-2 weeks after surgery
  Proportion of patients who achieve a pathological complete response following treatment

SECONDARY OUTCOMES:
Major pathological response (MPR) rates | 1-2 weeks after surgery
  The proportion of patients experiencing a major pathological response to neoadjuvant treatment.
Pathological tumor regression grade (TRG) | 1-2 weeks after surgery
  TRG is evaluated according to the AJCC system. TRG0-1 is defined as good response, TRG2 as moderate response, and TRG3 as poor response.
Rate of tumor down-staging | 1-2 weeks after surgery
  The proportion of patients experiencing tumor down-staging will be assessed by pathology.
Lymphocytes infiltration changes after treatment | 2 weeks before treatment and 1-2 weeks after surgery
  The categories, number and distribution of lymphocytes infiltrated in tumor and tumor stroma are measured by Multiplex immunofluorescence assay.
The expression of immune-related pathways | 2 weeks before treatment and 1-2 weeks after surgery
  The expression of immune-related pathways is measured by RNAseq.
Rectal MRI defined tumor regression | Baseline and 1 week before surgery
  Proportion of patients achieving rectal MRI-confirmed near or complete tumor regression.
Rectal MRI defined tumor down-staging | Baseline and 1 week before surgery
  Proportion of patients achieving rectal MRI-confirmed down-staging.
Rectal MRI defined tumor volume change | Baseline and 1 week before surgery
  The change of patients' tumor volume will be confirmed by rectal MRI.
Local recurrence(LR) rate | 3, 5 years
  Presence of adenocarcinoma within the rectal wall or within the mesorectum confirmed by pathology
Disease free survival (DFS) | 3, 5 years
  The three-year and five-year disease-free survival of patients.
Overall survival (OS) | 3, 5 years
  The three-year and five-year overall survival of patients.
Surgical complications | The surgical complications are assessed up to 5 years from the surgery
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc, which will also be assessed according to "Clavien-Dindo Classification of surgical complications".
R0 resection rate | Within two weeks after surgery
  Rate of complete tumor removal with negative microscopically resection margin.
Rate of sphincter-sparing surgery | Within two weeks after surgery
  Rate of sphincter-sparing surgery if surgery is performed.
Rate of adverse event | From date of randomization until the date of death from any cause, assessed up to 5 years
  Rate of adverse events will be assessed according to National Cancer Institution Common Terminology Criteria of Adverse Events (NCI-CTCAE) v.4.02. Adverse events of this trial will include immune-related adverse events, chemo- and radiotherapy related adverse events, and combined treatment-related adverse events.
Patient reported outcome: Quality of life according to questionnaire European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) (v 3.0) | Baseline and months 3, 6, 12, 24, 36, 60
  Score values from 1 (not at all) to 4 (very much) respectively from 1 (very poor) to 7 (excellent). Score outcome depends on score type.
Patient reported outcome: Quality of life according to questionnaire European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29) | Baseline and months 3, 6, 12, 24, 36, 60
  Score values from 1 (not at all) to 4 (very much). Score outcome depends on score type.
Patient reported outcome: Functional outcome according to Wexner score | Baseline and months 3, 6, 12, 24, 36, 60
  Five score values from "never" to "1 per day or more often". The more often the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiaolin Zhou, Ph.D, Study Chair — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No